CLINICAL TRIAL: NCT06898879
Title: Enhancing Veteran-Clinical Collaboration in VA Psychosocial Rehabilitation and Recovery Centers
Brief Title: Enhancing Veteran-Clinical Collaboration in VA PRRCs
Acronym: EVCC VPRRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5052-R; RX005052 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2025-03-12; First posted 2025-03-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Delusional Disorder; Bipolar Disorder; Major Depressive Disorder
Keywords: serious mental illness; psychosis; collaborative decision-making; shared decision-making; veterans; recovery; personal recovery; empowerment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid; Bipolar Disorder; Depressive Disorder, Major; Empowerment

STUDY DESIGN:
Intervention Model Description: The experimental design for this study is a 2-group randomized effectiveness trial, with assessments at baseline (month 0), post-intervention (month 3), and 3- and 6- post-intervention follow-ups (months 6 and 9). Veterans will be randomly assigned to either the CDST condition or to LU after completing baseline assessments. To maximize power for between-group comparisons, randomization will be 1:1 resulting in ~60 participants per group. Stratification may be introduced if necessary due to uneven or statistically different groups in key demographic domains (e.g., age, gender). Quantitative analyses will compare improvements in primary, secondary, and exploratory outcomes between the two groups, as described elsewhere. There are also qualitative outcomes associated with this study.
Who Masked: Outcomes Assessor
Masking Description: The research assistants who completes the assessments will be blind to condition, and will not attend any clinical team meetings or otherwise participate in any non-study related PRRC activities to maintain blindness. No study participants will be blinded. No other staff will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collaborative Decision Skills Training (Experimental): Collaborative Decision Skills Training (CDST) is the intervention group (experimental arm).
  Interventions: Behavioral: Collaborative Decision Skills Training
- Leveling Up (Active Comparator): Leveling Up is the active control arm.
  Interventions: Behavioral: Leveling Up

INTERVENTIONS:
Behavioral: Collaborative Decision Skills Training — An ten-session group-based skills training intervention that focuses on treatment-related decision-making in order to facilitate improved engagement in decision-making processes. CDST teaches assertiveness skills, problem solving, goal planning, and conflict negotiation, within the context of treatment planning and decision-making. Each session is 60 minutes long.
  Other Names: CDST
  Arms: Collaborative Decision Skills Training
Behavioral: Leveling Up — An ten-session group intervention that focuses on psychoeducation, befriending, and Veteran to Veteran support. Each session is 60 minutes long.
  Other Names: LU
  Arms: Leveling Up

SUMMARY:
Over 60% of Veterans with serious mental illness have a service-connected disability that impairs their ability to work, go to school, and/or have successful personal lives. Although traditional treatments tend to focus on symptom remission, Veterans prioritize a range of treatment goals, including personal empowerment and gaining personally meaningful skills. Increasing Veteran-clinician collaboration can help effectively align care with each Veteran's goals and support an empowering therapeutic experience. This project will evaluate the effectiveness of a group-based intervention intended to increase Veterans' comfort, confidence, knowledge, and skills to collaborate with their treatment teams. Findings from this study will contribute important knowledge about this intervention's effectiveness and how to enhance its effectiveness, especially for Veterans from minoritized groups. If the decision-making intervention is effective, it would help Veterans with serious mental illness, and might also help Veterans with other chronic health conditions, like PTSD and chronic pain.

DETAILED DESCRIPTION:
Recovery-oriented care is an imperative for the VA, particularly in mental health programming for Veterans with serious mental illness (SMI). Collaborative decision-making (CDM) is a recovery-oriented approach to treatment decision-making that supports meaningful involvement for patients across all aspects of decision- making, thereby empowering patients and facilitating better decision-making based on patient values, preferences, and cultural context. CDM is associated with several important outcomes including improved personal recovery, treatment engagement, treatment satisfaction, and social functioning. However, current levels of CDM among Veterans with SMI are low. Collaborative Decision Skills Training (CDST) is a promising 10-session group intervention that support Veterans to gain knowledge, skills, comfort, and confidence to collaborate with their clinicians and other members of their treatment teams. CDST has undergone initial testing in a VA Psychosocial Rehabilitation and Recovery Center (PRRC) and demonstrated feasibility for use among Veterans participating in PRRC care. This initial tests demonstrated preliminary evidence that CDST is effective at increasing Veteran-clinician collaboration, personal recovery, empowerment, treatment engagement, and social functioning.

Therefore, the proposed study will examine CDST's effectiveness among 119 Veterans with SMI participating in three PRRCs in the Southwestern United States (San Diego, Los Angeles, and Albuquerque). Veterans will be randomized to either CDST or active control (AC). The primary outcome measure will be functioning within the rehabilitation context, meaning Veteran CDM behavior during usual care VA mental health appointments. Secondary outcomes are treatment attendance, engagement, and satisfaction, along with functioning outside of the rehabilitation context (i.e., rehabilitation goal attainment, sense of personal recovery, empowerment symptom severity, and social functioning). Given that CDM is fundamentally an interaction between Veterans and their clinicians, the team will also assess whether clinician factors (i.e., engagement in CDST training or delivery; therapeutic alliance; work satisfaction; burnout; perceptions of self-efficacy; organizational climate; attitudes about recovery and CDM) moderate Veteran outcomes. Veterans in both groups will attend 10 hour- long group sessions held over 10 weeks.

All Veterans will complete an assessment battery at baseline, post-intervention, at three-month post- intervention follow-up, and at six-month follow-up. This will allow the team to assess durability of CDST's hypothesized benefits. Veterans who leave PRRC care and then return while the study is still active will complete one final assessment to further assess whether benefits are durable to re-entry to care. Additionally, the team will assess equity of benefits by assessing subgroup differences in benefits by race/ethnicity, gender, and sexual orientation. A team of Veterans and clinicians will be recruited to co-create consensus equity guidelines to support effective and equitable delivery of CDST in PRRCs.

The results of the proposed study will confirm CDST's benefits for Veterans in PRRC care and inform the utility of providing CDST broadly to Veterans with SMI. The results of this study will expand current understanding of CDM among Veterans with SMI by providing a large, diverse sample to 1) assess CDST's overall benefits; 2) durability and equity of those potential benefits; 3) whether and how clinician factors impact those potential benefits; and 4) identify how to deliver CDST and related interventions effectively and equitably.

ELIGIBILITY:
Inclusion Criteria:

1. be a Veteran currently receiving PRRC, MHICM and/or BHIP services at VA San Diego, Los Angeles, or Albuquerque (e.g., seen in the clinic in the past month or based on clinic criteria)
2. meet SAMHSA criteria of serious mental illness; i.e., "having (within the past year) a diagnosable mental, behavior, or emotional disorder that causes serious functional impairment that substantially interferes with or limits one or more major life activities," based on chart review and clinician consultation if needed
3. Be age 18 or above
4. Be fluent and literate in English.
5. Agree to have a subset of VA mental health treatment appointments audiotaped

Exclusion Criteria:

1. primary substance use or organic neurological disorder diagnosis determined by chart review
2. are determined by clinician and/or study staff to be at significant risk of exacerbation of symptoms, suicidal ideation, or other risk due to study participation
3. have a history and/or current risk of violence that clinicians and/or study staff determine to be too high risk to manage effectively in the study setting (e.g., poses a risk to Veterans or study staff).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-03 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Shared Decision-Making Coding System | Baseline to 3-month follow-up
  The Shared Decision-Making Coding System (SDM-CS) is a validated method of coding collaborative behaviors during treatment decision-making among patients with SMI and their providers. The SDM-CDS codes 9 elements of the decision process including goal setting, exploration of patient preference, and treatment alternatives. Coding for this measure is completed by recording frequency of specific interactions (e.g., the patient states a preference). Scores range from 0-18, where higher scores are better (indicating more collaborative behaviors).
Shared Decision-Making Coding System | Baseline to 6-month follow-up
  The Shared Decision-Making Coding System (SDM-CS) is a validated method of coding collaborative behaviors during treatment decision-making among patients with SMI and their providers. The SDM-CDS codes 9 elements of the decision process including goal setting, exploration of patient preference, and treatment alternatives. Coding for this measure is completed by recording frequency of specific interactions (e.g., the patient states a preference). Scores range from 0-18, where higher scores are better (indicating more collaborative behaviors).
Consumer-Created Opportunities for Active Involvement Coding System | Baseline to 3-month follow-up
  A validated measure for adults with SMI that codes presence of consumer driven collaborative behaviors, including sharing opinions about treatment effectiveness, making requests, and reflecting on the therapeutic relationship. This measure codes behaviors, so the minimum score is 0, and it has no maximum. Higher scores indicate more collaborative behaviors initiated by the consumer.
Consumer-Created Opportunities for Active Involvement Coding System | Baseline to 6-month follow-up
  A validated measure for adults with SMI that codes presence of consumer driven collaborative behaviors, including sharing opinions about treatment effectiveness, making requests, and reflecting on the therapeutic relationship. This measure codes behaviors, so the minimum score is 0, and it has no maximum. Higher scores indicate more collaborative behaviors initiated by the consumer.

SECONDARY OUTCOMES:
Singh O'Brien Level of Engagement Scale | Baseline to 3-month follow-up
  A 14-item clinician-rated measure using a 4-point Likert scale. Scores range from 0-42, where higher scores indicate more service engagement.
Singh O'Brien Level of Engagement Scale | Baseline to 6-month follow-up
  A 14-item clinician-rated measure using a 4-point Likert scale. Scores range from 0-42, where higher scores indicate more service engagement.
Client Satisfaction Questionnaire | Baseline to 3-month follow-up
  An 8-item self-report measure of client satisfaction, with scores ranging from 8-32. Higher scores indicate higher levels of satisfaction.
Client Satisfaction Questionnaire | Baseline to 6-month follow-up
  An 8-item self-report measure of client satisfaction, with scores ranging from 8-32. Higher scores indicate higher levels of satisfaction.
Canadian Occupational Performance Measure- Performance subscale | Baseline to 3-month follow-up
  A short interview-based measure that assesses goal attainment in a range of functional areas. In this study, the investigators will use the performance subscale. The performance subscale is rated between 1-10, where higher scores indicate better performance.
Canadian Occupational Performance Measure- Performance subscale | Baseline to 6-month follow-up
  A short interview-based measure that assesses goal attainment in a range of functional areas. In this study, the investigators will use the performance subscale. The performance subscale is rated between 1-10, where higher scores indicate better performance.
Goal Attainment Scaling | Baseline to 3-month follow-up
  An algorithm that identifies goals and goal attainment. Scores range from -2 to +2, with 0 meaning that the expected outcome was achieved, while lower scores mean that less favorable outcomes occurred, and higher scores mean that better than expected outcomes occurred.
Goal Attainment Scaling | Baseline to 6-month follow-up
  An algorithm that identifies goals and goal attainment. Scores range from -2 to +2, with 0 meaning that the expected outcome was achieved, while lower scores mean that less favorable outcomes occurred, and higher scores mean that better than expected outcomes occurred.
Maryland Assessment of Recovery in Serious Mental Illness | Baseline to 3-month follow-up
  A 25-item self-report measure that assesses personal alignment with six primary domains of recovery: self-direction or empowerment, holistic, nonlinear, strengths based, responsibility, and hope. Scores range from 25-125, with higher scores indicating higher levels of personal recovery.
Maryland Assessment of Recovery in Serious Mental Illness | Baseline to 6-month follow-up
  A 25-item self-report measure that assesses personal alignment with six primary domains of recovery: self-direction or empowerment, holistic, nonlinear, strengths based, responsibility, and hope. Scores range from 25-125, with higher scores indicating higher levels of personal recovery.
Personal and Social Performance scale | Baseline to 3-month follow-up
  A clinician-reported scale of patient ability in four areas: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. Scores range from 1-100, with higher scores indicating better social functioning.
Personal and Social Performance scale | Baseline to 6-month follow-up
  A clinician-reported scale of patient ability in four areas: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. Scores range from 1-100, with higher scores indicating better social functioning.
Shared Decision Making Questionnaire for Mental Health | Baseline to 3-month follow-up
  9 item measure of involvement in treatment decisions. Scores range from 0-45, with higher scores indicating high levels of involvement in treatment decisions.
Shared Decision Making Questionnaire for Mental Health | Baseline to 6-month follow-up
  9 item measure of involvement in treatment decisions. Scores range from 0-45, with higher scores indicating high levels of involvement in treatment decisions.
Problem-Solving Decision-Making Scale for Mental Health | Baseline to 3-month follow-up
  Self-report about preferences for involvement in treatment decision-making based on three brief vignettes. There are 18 items and a total score range from 18-90, with lower scores indicating preference for paternalistic (provider-determined) decision-making, higher scores indicating preference for self-determination in treatment decisions, and middle scores indicating preference for provider-self collaboration.
Problem-Solving Decision-Making Scale for Mental Health | Baseline to 6-month follow-up
  Self-report about preferences for involvement in treatment decision-making based on three brief vignettes. There are 18 items and a total score range from 18-90, with lower scores indicating preference for paternalistic (provider-determined) decision-making, higher scores indicating preference for self-determination in treatment decisions, and middle scores indicating preference for provider-self collaboration.
Patient Perceived Involved in Care Scale | Baseline to 3-month follow-up
  13 item self report measure. Scores range 0-13, with higher scores indicating higher perceived involvement in care.
Patient Perceived Involved in Care Scale | Baseline to 6-month follow-up
  13 item self report measure. Scores range 0-13, with higher scores indicating higher perceived involvement in care.
Empowerment Scale | Baseline to 3-month follow-up
  28 item self-report measure. Scores range from 0-112, where lower scores indicate more empowerment. Developed specifically for people with serious mental illness.
Empowerment Scale | Baseline to 6-month follow-up
  28 item self-report measure. Scores range from 0-112, where lower scores indicate more empowerment. Developed specifically for people with serious mental illness.
Behaviour and Symptom Identification Scale (BASIS) | Baseline to 3-month follow-up
  24 item self-report scale of broad mental health symptom severity, where higher scores indicate higher symptom severity. Total scores and subscales are based on weighted means of items, ranging of 0-4.
Behaviour and Symptom Identification Scale (BASIS) | Baseline to 6-month follow-up
  24 item self-report scale of broad mental health symptom severity, where higher scores indicate higher symptom severity. Total scores and subscales are based on weighted means of items, ranging of 0-4.
Clinical Global Impression | Baseline to 3-month follow-up
  Two item clinician rating of global illness severity. Higher scores indicate greater overall severity. Items are scored separately and both are on a 1-7 likert scale.
Clinical Global Impression | Baseline to 6-month follow-up
  Two item clinician rating of global illness severity. Higher scores indicate greater overall severity. Items are scored separately and both are on a 1-7 likert scale.
Brief Inventory of Psychosocial Functioning | Baseline to 3-month follow-up
  7 item self report measure of social functioning. Developed specifically for adults with serious mental illness. Total scores result in a 0-100 range where higher scores indicate higher functional impairment.
Brief Inventory of Psychosocial Functioning | Baseline to 6-month follow-up
  7 item self report measure of social functioning. Developed specifically for adults with serious mental illness. Total scores result in a 0-100 range where higher scores indicate higher functional impairment.

OTHER OUTCOMES:
Scale to Assess Therapeutic Relationship (patient and clinician versions) | Baseline to 3-month follow-up
  12 item measure to assess therapeutic alliance. One is patient-completed and one is clinician-completed. Total scores range from 0-48, where higher scores indicate higher therapeutic alliance.
Scale to Assess Therapeutic Relationship (patient and clinician versions) | Baseline to 6-month follow-up
  12 item measure to assess therapeutic alliance. One is patient-completed and one is clinician-completed. Total scores range from 0-48, where higher scores indicate higher therapeutic alliance.
Maslach Burnout Inventory | Every three months for 2.5 year clinical trial duration
  22 item measure of burnout. Includes three subscales, emotional exhaustion (9 items, total score ranging 0-54), depersonalization (5 items, total score ranging 0 - 30), and personal accomplishment (8 items, total score ranging from 0 -48). Total score therefore ranges from 0- 132. Higher scores indicate more burnout.
General Self-Efficacy Scale | Every three months for 2.5 year clinical trial duration
  10 item self report measure. Scores range from 10-40 with higher scores indicate higher self efficacy.
Recovery Knowledge Inventory | Every three months for 2.5 year clinical trial duration
  20 item clinical report measure. Scores range from 20-100 where higher scores indicate greater knowledge of recovery and stronger recovery orientation.
Task and Relational Climate Scale | Every three months for 2.5 year clinical trial duration
  six item self report scale of work climate related to two subconstructs (tasks and relationships with colleagues). Scoring ranges from 0-15 on each subscale and 0-30 overall, where higher scores indicate more positive climate.
Collaborative Decision Making Attitudes Measure | Every three months for 2.5 year clinical trial duration
  8 item clinician report measure. Scores range from 0-40 where higher scores indicate greater use of collaborative decision-making and greater alignment with collaborative decision-making as a clinical practice.
Work satisfaction | Every three months for 2.5 year clinical trial duration
  Single 10-point item (Overall, how satisfied are you with your current job?")
Perceived Cultural Competency | Baseline to 3-month follow-up
  9 item patient completed scale. Total scores range from 9-63 where higher scores indicate better cultural competency experiences with clinicians.
Perceived Cultural Competency | Baseline to 6-month follow-up
  9 item patient completed scale. Total scores range from 9-63 where higher scores indicate better cultural competency experiences with clinicians.
Qualitative interviews | Baseline to six month follow up
  Veteran semi-structured interviews focused on constructs aligned with quantitative outcomes including involvement in decision-making, treatment engagement, motivation, and satisfaction, and attainment of recovery goals. These interviews capture both primary, secondary, and pre-specified outcomes and will be triangulated with quantitative measures during the mixed methods integration process.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Treichler, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (3):
- United States (3):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying results in a publication will be shared. Deidentified data sets will be used for analysis and only these de-identified sets will be shared. All HIPAA identifiers, combinations of variables that might be used for re-identification, and proprietary information will be excluded. Audio data will not be shared; de-identified transcriptions and coding based on audio data will be. Only data needed to fulfill a requester's stated purpose will be shared. Therefore this plan will protect personal privacy of research subjects, prevent loss of confidentiality, and ensure the secure maintenance of propriety data and information.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be available six months after publication, and remain available for five years.
Access Criteria: Data will be shared with researchers and consumer advocates who provide a rationale and methodological sound plan for their use of the data. Acceptable uses include meta-analysis and mega-analysis, among other uses. Data sets provided to requesters will include data necessary for the requester's stated purpose, as long as the requester's purpose does not violate participant privacy, research ethics, or similar procedures.
  Requests for access must be made in writing including an explicit assurance that the recipient will not attempt to identify or re-identify any individual. Requests must be signed by a requester currently residing in the United States. The request must reference the publication or other source motivating the request along with the detailed purpose for the request. Requests should be made to the corresponding author or the principal investigator, but can be made to the Associate Chief of Staff for Research.